CLINICAL TRIAL: NCT01613196
Title: Evaluation of Positron Emission Tomography in Extrapulmonary Tuberculosis
Brief Title: Positron Emission Tomography in Extrapulmonary Tuberculosis
Acronym: TUBOGTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOM 11080; 2011-A01658-33 (Other: IDRCB)
Record Dates: First submitted 2012-05-14; First posted 2012-06-07 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Extrapulmonary Tuberculosis; Lymph Node Tuberculosis; Bone Tuberculosis
Keywords: Extrapulmonary tuberculosis; FDG-TEP; cohorts
MeSH Terms: conditions — Tuberculosis, Extrapulmonary; Tuberculosis, Lymph Node; Tuberculosis, Osteoarticular | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Positron Emission Tomography (Experimental): Positron Emission Tomography
  Interventions: Other: Positron Emission Tomography with 18F-Fluoro-deoxy-glucose

INTERVENTIONS:
Other: Positron Emission Tomography with 18F-Fluoro-deoxy-glucose — 2 or 3 FDG-PET scans will be performed in all patients : at inclusion*, end of treatment and 6 months after completion of treatment in cases of persistent uptake
  *except if already done in the last 15 days.
  Other Names: PET with 18 FDG

SUMMARY:
Tuberculosis (TB) remains a major public health problem. In extra-pulmonary forms, evidence of bacteriological cure is difficult to be obtained raising the need for other therapeutic assessment tools. 18F-Fluoro-deoxy-glucose (FDG) is a glucose analogue widely used in Positron Emission Tomography (PET). Its uptake is high in cancer cells and in inflammatory cells, especially in active TB foci. The hypothesis is a decrease in the uptake of FDG in the foci of TB during treatment permitting a non-invasive monitoring of therapeutic response. The main objective is to describe the evolution under treatment of the FDG uptake in PET imaging in TB foci in patients cured from lymph node and bone TB. Secondary objectives are to compare the decrease of FDG uptake according to type of location, to define the frequency of localizations revealed by FDG-PET and their impact on therapeutic management at the beginning and the end of treatment, and to describe the evolution of PET in patients not cured.

DETAILED DESCRIPTION:
Longitudinal observational multicenter pilot study. 55 patients to be included Total duration of the study: 51 months. Inclusion period: 27 months Follow up period: 18 to 24 months Number of participating centers: 11 Average number of inclusion per month per center: 1-2

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Affiliated to a social security system or "AME"
* Patient informed of the objectives and constraints of the study and giving informed consent
* Patient can keep lying valid at least 30 minutes
* Patient not HIV infected or, if infected, with CD4 counts> 200/mm3 for at least 3 months

Exclusion Criteria:

* Suspicion of other concurrent infection
* Severe immunosuppression in case of HIV infection
* Inflammatory disease
* Pregnant or nursing women
* Radiation therapy
* Uncontrolled diabetes
* Prolonged corticosteroid therapy (> 20mg/day)
* Patient unable to sustain injected CT scan and MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
ΣSUVmax variations between the beginning and end of treatment and during follow-up post-treatment, in patients considered cured | 6 to 18 months
  To measure FDG uptake and evolution, the ΣSUVmax will be used. SUV ("Standard Uptake Value") is defined as tissue concentration of FDG / administered FDG dose / patient weight. ΣSUVmax is the sum of the maximum SUV measured in every TB foci. ΣSUVmax variations between the beginning and the end of treatment, and 6 months later in cases of persistent uptake at the end of treatment will be studied in patients considered cured

SECONDARY OUTCOMES:
Change in SUVmax differences in the lesions according to their location in cured patients. | 6 to 18 months
  SUV variations between the beginning and the end of treatment, and 6 months later in cases of persistent uptake at the end of treatment will be studied in the lesions according to their location in cured patients
Variations ΣSUVmax and SUVmax in individual lesions in patients not cured. | 6 to 18 months
  ΣSUVmax variations between the beginning and the end of treatment, and 6 months later in cases of persistent uptake at the end of treatment will be studied in patients not cured.
Frequency, type and consequences on the therapeutic management of lesions revealed by FDG-PET. | 6 to 18 months
  Changes in composition or treatment duration will be identified and reported to the information provided by FDG-PET during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yeni, MD, PHD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- BICHAT Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided